CLINICAL TRIAL: NCT00434421
Title: A Safety and Pilot Dosing Study for Sublingual-Oral Administration of Glycerinated German Cockroach Allergenic Extract in Pediatric and Adult Subjects With Cockroach Allergy and Perennial Allergic Rhinitis With or Without Asthma
Brief Title: Sublingual Cockroach Safety in Adults With Cockroach Allergy & Perennial Allergic Rhinitis With or Without Asthma
Acronym: SCSS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Inner-City Asthma Consortium (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DAIT ICAC-10
Record Dates: First submitted 2007-02-12; First posted 2007-02-13 (Estimated); Results first posted 2015-05-12 (Estimated); Last update posted 2015-06-11 (Estimated); Status verified 2015-06

CONDITIONS: Allergy; Asthma
Keywords: Perennial Allergic Rhinitis; Asthma; Sublingual Immunotherapy (SLIT)
MeSH Terms: conditions — Hypersensitivity; Asthma; Rhinitis, Allergic, Perennial

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- German Cockroach Allergen Dosing Group (Experimental): Glycerinated German Cockroach Allergenic Extract
  Interventions: Drug: Glycerinated German cockroach allergenic extract; Drug: Placebo

INTERVENTIONS:
Drug: Glycerinated German cockroach allergenic extract — Initially each subject underwent a 1-day, 8-dose escalation (e.g., one dose of placebo, 0.14 milliliters [mL], followed by 7 escalating doses of Glycerinated German Cockroach Allergenic Extract until the Maximum Study Dose [0.42 mL, 1:10 wt/vol] or Maximum Tolerated Dose was achieved). This maximum dose became the daily dose - maintenance dose- of Glycerinated German Cockroach Allergenic Extract for the following 14 days.The maintenance dose of 0.42 mL was calculated to contain 3685 bioequivalent allergy units (BAU), with approximately 4.2 mg of German cockroach allergen Bla g 2 and 50 mg of Bla g 1 per dose. Route of administration: sublingual-oral route.
  Other Names: Blattella germanica allergenic extract; Cockroach antigen (CR antigen)
Drug: Placebo — Placebo was administered only as the first dose (e.g., representing no Glycerinated German Cockroach bioequivalent allergy units) during the initial 1-day, 8-dose escalation, otherwise referred to as the Preliminary Dosing Visit. Refer to the Glycerinated German cockroach allergenic extract treatment for more details. Route of administration: sublingual-oral route.
  Other Names: Glycerinated German cockroach allergenic extract placebo

SUMMARY:
Immunotherapy may help reduce symptoms of allergy and asthma. Problems concerning compliance and adverse events with subcutaneous allergen immunotherapy have generated interest in delivering immunotherapy sublingually (under the tongue). The purpose of this study is to evaluate the safety of a cockroach extract given sublingually to people with perennial (year-round) allergic rhinitis, with or without asthma.

DETAILED DESCRIPTION:
The prevalence of asthma has dramatically increased in many parts of the world. Currently, there is no effective way to prevent development of allergic rhinitis and asthma and no cure. Sublingual immunotherapy (SLIT), a type of therapy in which allergens are placed under the tongue, may be a way to control and possibly prevent allergic rhinitis and asthma. However, detailed research of this approach is limited.

The purpose of this study is to evaluate the safety and tolerability of a sublingual cockroach extract given to people with perennial allergic rhinitis. Participants in this study will include people both with and without asthma.

Participation in this study will last a little more than 2 weeks. Participants will be stratified by age (oldest to youngest age group) and degree of cockroach sensitivity. Each age group will be enrolled after the previous group's safety data have been reviewed. At study entry (Day 0), participants will receive a dose of placebo and then up to seven incremental doses of cockroach extract at 15-minute intervals while observed by the clinic nurse. Doses will continue to be given until a sign or symptom occurs that indicates the participant is having difficulty tolerating the drug, or until the maximum study dose is reached.

At the Principal Investigator's discretion, participants who were able to achieve the maximum study dose will be invited to continue onto the 2-week treatment course of the study. These participants will return on Days 1 and 2 to the clinic to self-administer the maximum study dose of cockroach extract. After self-administering the maximum study dose, participants will be observed by the clinic nurse for 30 minutes. On Days 3 through 14, participants will take the maximum study dose of cockroach extract daily at home. Participants will be asked to keep a diary and record signs or symptoms experienced after taking each dose.

Skin tests, breathing tests, and blood collection will occur at study screening. At study entry, participants will be taught to use an EpiPen in the event of a severe allergic reaction at any time during the study. A physical exam/fitness assessment will be done at study screening, study entry, and the final visit. Unused extract will be collected at the final visit from participants who entered the 2-week treatment course of the study.

The reference for this study is SCSS (Sublingual Cockroach Safety Study) in the provided citation: Wood RA, Togias A, Wildfire J et al. Development of cockroach immunotherapy by the Inner-City Asthma Consortium. J Allergy Clin Immunol. 2014 Mar;133(3):846-52. PubMed ID: 24184147).

ELIGIBILITY:
Inclusion Criteria for All Participants:

* History of perennial allergic rhinitis with or without asthma for a minimum of 1 year prior to study entry
* Positive skin prick test to German cockroach performed along with negative (saline) and positive (histamine) controls
* Willing to sign EpiPen training form
* Parent or guardian willing to provide informed consent, if applicable

Inclusion Criteria for Participants with Asthma:

* Diagnosis of well-controlled, mild to moderate persistent asthma, defined as having symptoms at least 3 times a week with no controller medication OR less than 3 times a week on controller medication. More information about this criterion can be found in the protocol.
* Diagnosis of asthma made over 1 year prior to study entry

Exclusion Criteria:

* Have severe, persistent asthma (according to National Asthma Education and Prevention Program [NAEPP] classification) as evidenced by those who require a dose of greater than 500 mcg of fluticasone/day or equivalent of another inhaled corticosteroid OR who have been hospitalized for asthma within 6 months prior to study entry
* Life-threatening asthma exacerbation requiring intubation or mechanical ventilation or resulting in a hypoxic seizure in the 2 years prior to study entry
* History of anaphylaxis of Grade 2 or higher as defined in the protocol
* Unstable angina, significant arrhythmia, uncontrolled hypertension, or other chronic or immunologic diseases that, in the opinion of the investigator, may interfere with the study or pose additional risk to the patient. More information about this criterion can be found in the protocol.
* Taking medications that could induce gastrointestinal reactions during the study. Participants taking such medications must prove to be stable with no side effects for at least 3 months prior to study screening to be considered eligible.
* Received an investigational drug in the 30 days prior to study entry OR plan to receive an investigational drug during the study
* Received allergen immunotherapy in the 180 days prior to screening or plan to initiate or resume allergen immunotherapy during the study
* Taking tricyclic antidepressants or beta-adrenergic blocker drugs
* Received omalizumab in the 3 months prior to study screening
* Known contraindication to therapy with cockroach extract used in this study
* Mental illness that would interfere with the participant's ability to comply to study requirements
* History of drug or alcohol abuse that, in the opinion of the investigator, would interfere with the study
* Plan to leave study area during the study
* Does not primarily speak English, including caretakers of participants when the participant is a child
* Cannot perform spirometry
* Pregnant or breastfeeding

Ages: 5 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 28 (Actual)
Dates: Start 2007-02; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Wood, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University School of Medicine, 600 North Wolfe St, CMSC 1102, Baltimore, Maryland, United States

REFERENCES:
- [Background] Cox LS, Larenas Linnemann D, Nolte H, Weldon D, Finegold I, Nelson HS. Sublingual immunotherapy: a comprehensive review. J Allergy Clin Immunol. 2006 May;117(5):1021-35. doi: 10.1016/j.jaci.2006.02.040. PMID 16675328
- [Background] Gidaro GB, Marcucci F, Sensi L, Incorvaia C, Frati F, Ciprandi G. The safety of sublingual-swallow immunotherapy: an analysis of published studies. Clin Exp Allergy. 2005 May;35(5):565-71. doi: 10.1111/j.1365-2222.2005.02240.x. PMID 15898976
- [Background] Nelson HS. Advances in upper airway diseases and allergen immunotherapy. J Allergy Clin Immunol. 2006 May;117(5):1047-53. doi: 10.1016/j.jaci.2005.12.1306. Epub 2006 Mar 6. PMID 16675331
- [Background] Wilson DR, Lima MT, Durham SR. Sublingual immunotherapy for allergic rhinitis: systematic review and meta-analysis. Allergy. 2005 Jan;60(1):4-12. doi: 10.1111/j.1398-9995.2005.00699.x. PMID 15575924
- [Result] Wood RA, Togias A, Wildfire J, Visness CM, Matsui EC, Gruchalla R, Hershey G, Liu AH, O'Connor GT, Pongracic JA, Zoratti E, Little F, Granada M, Kennedy S, Durham SR, Shamji MH, Busse WW. Development of cockroach immunotherapy by the Inner-City Asthma Consortium. J Allergy Clin Immunol. 2014 Mar;133(3):846-52.e6. doi: 10.1016/j.jaci.2013.08.047. Epub 2013 Nov 1. PMID 24184147
- See also: National Institute of Allergy and Infectious Diseases (NIAID) — http://www.niaid.nih.gov/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The result tables represent the safety population: all subjects that initiated the 1-day, 8-dose escalation, otherwise referred to as the Preliminary Dosing Visit. One subject in the 8-17 age group withdrew from the study after this timepoint and was replaced with another participant.
Groups:
- German Cockroach Allergen Dosing Group: Initially each subject underwent a 1-day, 8-dose escalation (e.g., one dose of placebo, 0.14 milliliters [mL], followed by 7 escalating doses of Glycerinated German Cockroach Allergenic Extract until the Maximum Study Dose [0.42 mL, 1:10 wt/vol] or Maximum Tolerated Dose was achieved). This maximum dose became the daily dose - maintenance dose- of Glycerinated German Cockroach Allergenic Extract for the following 14 days.The maintenance dose of 0.42 mL was calculated to contain 3685 bioequivalent allergy units (BAU), with approximately 4.2 mg of German cockroach allergen Bla g 2 and 50 mg of Bla g 1 per dose. Route of administration: sublingual-oral route.
Period: Overall Study
Arm/Group | German Cockroach Allergen Dosing Group
Started | 28
Completed | 26
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — Non-compliance with study treatment | 1

BASELINE CHARACTERISTICS:
Population: All study participants who were initiated onto the initial placebo study treatment during the Preliminary Dosing Visit.
Arm/Group | German Cockroach Allergen Dosing Group
Number analyzed (Participants) | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 19
  Between 18 and 65 years | 9
  >=65 years | 0
Age, Customized [Number; unit: participants]
  18-55 years | 9
  8-17 years | 10
  5-7 years | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 28
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 22
  White | 3
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  United States | 28
German Cockroach Skin Test Sensitivity [Number; unit: participants] — Sensitivity to German cockroach allergen as measured by wheal size at baseline skin prick test. High sensitivity is defined as equal to or greater than a 6 mm wheal; low sensitivity, as equal to or greater than 3 mm wheal and less than 6 mm.
  participants
    High | 18
    Low | 10
Asthma status (Mild-to-moderate persistent asthma) [Number; unit: participants] — Asthma status as defined by self-reported doctor diagnosis over a year before study pre-screening and reported symptoms and controller medication use. Mild-to-moderate persistent asthma is defined as (i) symptoms at least 3 times a week on no controller medication or (ii) symptoms < 3 times a week on controller medication. Qualifying controller medication regimens included: leukotriene; fluticasone (up to 500 mcg/day) or equivalent; leukotriene modifier plus fluticasone (up to 500 mcg/day) or equivalent; salmeterol plus fluticasone (up to 500 mcg/day) or equivalent.
  participants
    Yes | 10
    No | 18

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants Who Discontinue Study
Description: Proportion of participants who discontinued study for any reason following initiation of treatment (any participant who receives the initial placebo dose will be considered initiated onto treatment)
Time Frame: Initial placebo dose to end of 2-week treatment course (maximum study dose)
Population: Safety Population: All study participants who were initiated onto the initial placebo study
Measure: Number; unit: Percentage of Participants
Arm/Group | German Cockroach Allergen Dosing Group
Number analyzed (Participants) | 28
Percentage of Participants | 7.1

ADVERSE EVENTS:
Time Frame: Initial placebo dose to end of 2-week treatment course
Arm/Group | German Cockroach Allergen Dosing Group
Serious Adverse Events (participants affected / at risk) | 0/28
Other Adverse Events (participants affected / at risk) | 15/28
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | German Cockroach Allergen Dosing Group (N=28)
EAR PRURITUS (Ear and labyrinth disorders) | 3 (3)
EYE PRURITUS (Eye disorders) | 2 (2)
CRAMPS (Gastrointestinal disorders) | 1 (1)
DIARRHEA (Gastrointestinal disorders) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 1 (1)
SALIVARY HYPERSECRETION (Gastrointestinal disorders) | 1 (1)
VOMITING (Gastrointestinal disorders) | 1 (1)
CHEST DISCOMFORT (Respiratory, thoracic and mediastinal disorders) | 3 (3)
COUGH (Respiratory, thoracic and mediastinal disorders) | 2 (2)
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 1 (1)
NASAL DISCOMFORT (Respiratory, thoracic and mediastinal disorders) | 1 (1)
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 2 (2)
SHORTNESS OF BREATH (Respiratory, thoracic and mediastinal disorders) | 1 (1)
SNEEZING (Respiratory, thoracic and mediastinal disorders) | 1 (1)
THROAT IRRITATION (Respiratory, thoracic and mediastinal disorders) | 6 (8)
WHEEZING (Respiratory, thoracic and mediastinal disorders) | 1 (1)
ERYTHEMA (Skin and subcutaneous tissue disorders) | 1 (1)
ORAL PRURITUS (Skin and subcutaneous tissue disorders) | 5 (5)
PRURITUS (Skin and subcutaneous tissue disorders) | 3 (4)
RASH (Skin and subcutaneous tissue disorders) | 4 (4)
RASH PRURITIC (Skin and subcutaneous tissue disorders) | 1 (1)
URTICARIA (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No